CLINICAL TRIAL: NCT06613659
Title: Cohort Study on the Efficacy of Traditional Chinese Medicine Syndrome Differentiation Scheme in Adjuvant Treatment of Severe Pneumonia Based on the Real World
Brief Title: Cohort Study on the Treatment of Severe Pneumonia with Traditional Chinese Medicine
Status: Not yet recruiting | Type: Observational
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: RESEARCH-SEVERE PNEUMONIA
Record Dates: First submitted 2024-09-21; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2023-11

CONDITIONS: Community-Acquired Infections
Keywords: Community-Acquired Infections; Traditional Chinese Medicine; Cohort study
MeSH Terms: conditions — Community-Acquired Infections | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treatment cohort of integrated traditional Chinese and Western Medicine: Taking the use of traditional Chinese medicine syndrome differentiation treatment as the exposure factor, the continuous use of traditional Chinese medicine for 3-5 days was defined as mild exposure, continuous use of traditional Chinese medicine for 6-10 days as moderate exposure, and continuous use of traditional Chinese medicine for more than 10 days as severe exposure. The exposure group was treated with syndrome differentiation of traditional Chinese medicine combined with conventional Western Medicine (treatment cohort of integrated traditional Chinese and Western Medicine).
  Interventions: Drug: traditional Chinese medicine (TCM)
- Western medicine treatment queue: The non exposure group (Western medicine treatment cohort) used conventional western medicine treatment but not standardized TCM syndrome differentiation treatment.
  Interventions: Drug: non traditional Chinese medicine (non-TCM)

INTERVENTIONS:
Drug: traditional Chinese medicine (TCM) — Taking the use of traditional Chinese medicine syndrome differentiation treatment as the exposure factor, the continuous use of traditional Chinese medicine for 3-5 days was defined as mild exposure, continuous use of traditional Chinese medicine for 6-10 days as moderate exposure, and continuous use of traditional Chinese medicine for more than 10 days as severe exposure. The exposed group used TCM syndrome differentiation therapy combined with conventional western medicine treatment (integrative medicine treatment cohort), and the non exposed group used conventional western medicine treatment without standardized TCM syndrome differentiation treatment (Western medicine treatment cohort). The treatment plan was formulated by the clinician, and the researcher did not intervene.
  Groups: Treatment cohort of integrated traditional Chinese and Western Medicine
Drug: non traditional Chinese medicine (non-TCM) — Taking the use of traditional Chinese medicine syndrome differentiation treatment as the exposure factor, the continuous use of traditional Chinese medicine for 3-5 days was defined as mild exposure, continuous use of traditional Chinese medicine for 6-10 days as moderate exposure, and continuous use of traditional Chinese medicine for more than 10 days as severe exposure. The exposed group used TCM syndrome differentiation therapy combined with conventional western medicine treatment (integrative medicine treatment cohort), and the non exposed group used conventional western medicine treatment without standardized TCM syndrome differentiation treatment (Western medicine treatment cohort). The treatment plan was formulated by the clinician, and the researcher did not intervene.
  Groups: Western medicine treatment queue

SUMMARY:
This is a multicenter, prospective cohort study, with syndrome differentiation and treatment of traditional Chinese medicine as the exposure factor. Patients using syndrome differentiation of traditional Chinese medicine combined with conventional treatment of Western medicine are classified as the treatment cohort of Integrated Chinese and Western medicine, and patients using conventional treatment of Western medicine only are classified as the treatment cohort of Western medicine

DETAILED DESCRIPTION:
Severe pneumonia is a severe respiratory disease with high mortality, many complications and poor prognosis. Traditional Chinese medicine has certain curative effect in the adjuvant treatment of severe pneumonia, but there is a lack of systematic TCM syndrome differentiation scheme and its curative effect evaluation in the real medical environment. The cohort study on the efficacy of TCM syndrome differentiation scheme in the adjuvant treatment of severe pneumonia is conducive to providing new evidence for the optimization and evidence-based evaluation of TCM treatment scheme for severe pneumonia. Therefore, this study took severe pneumonia as the research object, standardized use of traditional Chinese medicine diagnosis and treatment scheme as the exposure factor, carried out a multi center prospective cohort study, used the 90 day mortality, 28 day mortality, treatment failure rate, etc., to evaluate the clinical efficacy and safety of integrated traditional Chinese and Western medicine in the treatment of severe pneumonia, and provided evidence for the application and promotion of traditional Chinese medicine in severe pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* It met the diagnostic criteria of severe pneumonia;
* Age ≥ 18 years old, regardless of gender.
* Voluntary treatment.
* Sign the informed consent form.

Exclusion Criteria:

* Pregnant or lactating women;
* Patients with mental illness who are unable to cooperate or unwilling to cooperate with follow-up;
* Those who are participating in clinical trials of other drugs;
* Known allergic to therapeutic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe community-acquired pneumonia (CAP) is a severe respiratory disease with further development and deterioration of lung tissue inflammation, causing organ dysfunction and even life-threatening. Patients with SCAP are prone to hypoxemia, respiratory failure, septic shock, leading to multiple organ failure and poor prognosis. Western medicine treatment of SCAP mainly focuses on anti infection and mechanical ventilation. Although new intervention measures and management concepts are constantly optimized, the mortality rate of SCAP is still high. The treatment of SCAP is facing a severe situation, so it is necessary to seek new adjuvant therapy.
Sampling Method: Probability Sample
Enrollment: 1016 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
90-day mortality | Mortality on the 90th day of treatment
  Calculate the proportion of patients who died of the disease on the 90th day of treatment

SECONDARY OUTCOMES:
28-day mortality | Calculate the proportion of patients who died of the disease on the 28th day after discharge
treatment failure rate | Early treatment failure was defined as clinical deterioration within 72 hours of treatment. Late treatment failure between 72 hours and to 28 days.
  The primary efficacy outcome was the rate of treatment failure, which includes treatment failure that occurred early,late, or at both times.
time to clinical stability | every day in the treatment.
  temperature of 37.2°C orlower, heart rate of 100 beats/min or lower, systolic blood pressure of 90 mm Hg or higher, and arterial oxygen tension of 60 mm Hg or higher when the patient was not receiving supplemental oxygen.
ICU stay time | the 28 days of the treatment phase.
  length of ICU and hospital stays will be recorded.
hospitalization time | the 28 days of the treatment phase
  length of hospital stays will be recorded.
Mechanical ventilation time | the 28 days of the treatment phase
  Time of invasive mechanical ventilation
SOFA score | The sofa scores of the first, seventh, fourteenth, twenty-first and twenty-eight days of admission and the first, second and third months after discharge were counted.
  Sequential Organ Failure Assessment.It is a scoring system for evaluating and monitoring the organ function of critically ill patients.The minimum score is 0 and the maximum is 24. The higher the score, the worse the result.
Quality of life | The scores of the first, seventh, fourteenth, twenty-first and twenty-eight days of admission and the first, second and third months after discharge were counted
  Score according to the quality of life table,the minimum score is 12 points, and the maximum score is 60 points. The higher the score, the worse the result.
TCM syndrome score | The TCM syndrome scores of the first, seventh, fourteenth, twenty-first and twenty-eight days and the first, second and third months after discharge were counted
  Traditional Chinese Medicine Syndrome Points.Including cough, expectoration, dyspnea, chest pain, anorexia and fatigue, each item is rated as 1-5 points from mild to severe.The minimum score is 6 points and the maximum score is 30 points. The higher the score, the worse the result.
90 day readmission rate | The proportion of rehospitalization due to exacerbation within 90 days after discharge was recorded
  The proportion of rehospitalization due to exacerbation within 90 days after discharge was recorded

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan, China